CLINICAL TRIAL: NCT06932770
Title: Anti-aging Efficacy Study With Food Supplement and Cosmetic Routine vs Placebo
Brief Title: Anti-aging Efficacy of Food Supplement and Cosmetic Routine
Acronym: In&Out
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: SGS proderm GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 25.0036-23
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Aging; Wrinkle

STUDY DESIGN:
Intervention Model Description: Split-face design. Subjects will be divided equally in 2 treatment groups (food supplement active or food supplement placebo). Group 1 will receive treatments A and B (food supplement active with cosmetic active on one volar forearm and one side of face and cosmetic placebo on the other volar forearm and side of face) and group 2 C and D (food supplement placebo with cosmetic active on one volar forearm and one side of face and cosmetic placebo on the other volar forearm and side of face). Treatments will be randomly and balanced assigned to left and right test area in each group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Food supplement and cosmetic routine (Experimental): The "food supplement and cosmetic routine" arm will consume the food supplement active and apply the skin care product active.
  Interventions: Dietary Supplement: Food Supplement active; Other: Skin care product active
- Food supplement (Experimental): The "food supplement" arm will consume the food supplement active and apply the skin care product placebo.
  Interventions: Dietary Supplement: Food Supplement active; Other: Skin care product placebo
- Cosmetic routine (Experimental): The "cosmetic routine" arm will consume the food supplement placebo and apply the skin care product active.
  Interventions: Dietary Supplement: Food supplement placebo; Other: Skin care product active
- Placebo (Placebo Comparator): The "placebo" arm will consume the food supplement placebo and apply the skin care product placebo.
  Interventions: Dietary Supplement: Food supplement placebo; Other: Skin care product placebo

INTERVENTIONS:
Dietary Supplement: Food Supplement active — The food supplement active (2 soft gels) will be consumed once per day with a large glass of water.
  Arms: Food supplement; Food supplement and cosmetic routine
Dietary Supplement: Food supplement placebo — The food supplement placebo (2 soft gels) will be consumed once per day with a large glass of water.
  Arms: Cosmetic routine; Placebo
Other: Skin care product active — The cosmetic skin care product active will be applied twice daily to half of the face and to one volar forearm.
  Arms: Cosmetic routine; Food supplement and cosmetic routine
Other: Skin care product placebo — The cosmetic skin care product placebo will be applied twice daily to half of the face and to one volar forearm.
  Arms: Food supplement; Placebo

SUMMARY:
The aim of this study is to investigate the impact of a topical and an oral product alone and in combination compared to placebo on skin aging

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female
* From 40 to 70 years of age, in order to include sufficient subjects for the study, if necessary, the age may be gradually increased to 70 years or decreased to 40 years
* Healthy skin in the test areas
* Visible wrinkles in the face (grade 3 to 6 according to proderm wrinkle score)

For biopsy subpanel:

- Vaccination of tetanus within the last 10 years

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Active skin disease at the test area
* Documented allergies to face/eye care products and food supplements or their ingredients
* Intake of dietary supplements within the last 3 months before the start of the study
* Diabetes mellitus
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension (if not adjusted with medication), cardiovascular diseases
* Epilepsy
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, freckles, etc. at the test area that could influence the investigation
* Regular use of tanning beds
* Any topical medication at the test area within the last 3 days prior to the start of the study
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) and/or within the last 7 days prior to the start of the study
* Therapy with antibiotics within the last 2 weeks prior to the start of the study
* Past cosmetic surgery procedure in the test area (e.g. laser, facelift)
* Cosmetic surgery procedure in the test area, e.g. IPL (Intensed Pulsed Light), botox, chemical peel, dermabrasion within the last 2 years prior to the start of the study and/or throughout the entire course of the study
* Medical treatment for wrinkle reduction (e.g. peeling with vitamin A or fruit acids) on the face within the last 2 weeks prior to the start of the study

For biopsy subpanel:

* Regular medication with anti-coagulating drugs like Aspirin®, Macumar®, etc. (e.g. for thrombosis prophylaxis) within up to 15 days prior to the taking of the biopsies
* History of complications at wound healing (e.g. keloids, hypertrophic scars or contracture scar)
* Known intolerance to local anaesthetics
* Known Sensitivity to any dressing systems

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Anti-wrinkle efficacy | 12 weeks
  Change from baseline in anti-wrinkles efficacy (assessed on three-dimensional structure of the wrinkles in the periorbital regions) after 6 and 12 weeks. Anti-wrinkle efficacy will be assessed using DermaTOP. Parameters measured: Rz and Ra, representing mainly the rough structure (Rz) or the finer skin structure (Ra).

SECONDARY OUTCOMES:
Skin barrier function | 12 weeks
  Change from baseline in skin barrier function (assessed onTransepidermal water loss (TEWL) by Tewameter [g/(m²h)]) after 6 and 12 weeks
Skin hydration | 12 weeks
  Change from baseline in skin hydration (assessed on skin capacitance by Corneometer) after 6 and 12 weeks
Skin firmness | 12 weeks
  Change from baseline in skin firmness (assessed by R0 (Uf) by Cutometer [mm]) after 6 and 12 weeks
Skin elasticity | 12 weeks
  Change from baseline in skin elasticity (assessed by R7 (Ur/Uf) by Cutometer) after 6 and 12 weeks
Wrinkles and fine lines | 12 weeks
  Change from baseline for wrinkles and fine lines (assessed on VISIA-CR Image analysis) after 6 and 12 weeks
Skin aging hallmarks | 12 weeks
  Change from baseline in skin hallmarks of aging (assessed on 3mm punch skin biopsies) after 12 weeks in a subpanel of participants
Product traits | 12 weeks
  Subjective evaluation of product traits assessed via questionnaire after 6 and 12 weeks.
  Product traits will be assessed by the subjects with a list of closed questions with the following predefined identical options to tick:
  * 2 = Fully disagree;
  * 1 = Rather disagree;
    1. = Rather agree;
    2. = Fully agree

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Unbereit, Principal Investigator — SGS proderm GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No